CLINICAL TRIAL: NCT04066504
Title: A Non-interventional, Multi-national, Multi-center Post-authorization Safety Study (PASS) to Assess the Long Term Safety and Tolerability of Odomzo (Sonidegib) Administered in Patients With Locally Advanced Cell Carcinoma (laBCC)
Brief Title: Post-authorization Safety Study on the Long Term Safety of Sonidegib in Patients With Locally Advanced Cell Carcinoma
Acronym: NISSO
Status: Completed | Type: Observational
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CLDE225A2404
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Basal Cell Carcinoma
Keywords: locally advanced basal cell carcinoma; laBCC
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — sonidegib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Sonidegib: Patients with laBCC undergoing sonidegib treatment in routine clinical practice
  Interventions: Drug: sonidegib

INTERVENTIONS:
Drug: sonidegib — Sonidegib 200 mg orally taken once daily (dose modifications according to the approved local country prescribing information are permitted)
  Other Names: LDE225

SUMMARY:
Collect real world safety data on the use of sonidegib in adult patients with laBCC. Document major safety parameters such as on treatment deaths, adverse events (AEs)/ serious adverse events (SAEs) and discontinuation secondary to AEs.

DETAILED DESCRIPTION:
This is a non-interventional, multinational, multi-center post-authorization safety study (PASS), to assess the safety of sonidegib administered in routine clinical practice in patients with laBCC who are not amendable to curative surgery or radiation therapy. This study is observational in nature and does not impose a therapy protocol, diagnostic/therapeutic interventions or a specific visit schedule. For this study, each enrolled patient will be followed up for 3 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or equivalent document (e.g., written information) as per country regulation
* Patients aged 18 years or older with a diagnosis of laBCC who are not amenable to curative surgery or radiation therapy
* Patients must be treated with sonidegib 200 mg orally taken once daily (dose modifications according to the approved local country prescribing information are permitted)
* Sonidegib treatment must be started either at the first visit for this study or prior to study entry.

Exclusion Criteria:

* Patients treated with any hedgehog pathway inhibitor besides sonidegib within 3 months prior to study entry
* Patients currently enrolled in an interventional clinical trial
* Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of the Summary of Product Characteristics (SmPC)
* Pregnancy and breast-feeding
* Women of childbearing potential who do not comply with the Odomzo Pregnancy Prevention Programme (as defined in sections 4.4 and 4.6 of the approved SmPC).
* Male patients who are unable to follow or comply with the required contraception measures (as defined in sections 4.4 and 4.6 of the approved SmPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with laBCC undergoing treatment with sonidegib.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with AEs/SAEs | 3 years
  including on-treatment deaths and discontinuation due to AEs/SAEs

SECONDARY OUTCOMES:
Proportion of patients with AEs of special interest (AESI) or populations | 3 years
  in patients with: relevant polymorphism, ≥65 yrs, hepatic or renal impairment, female patients with child bearing potential using anticonceptives, anemia (hemoglobin <9 g/dL), recent myocardial ischemia or cardiac failure, concomitant medications with known risk of creatine kinase elevation

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Gutzmer, Principal Investigator — Universitätsklinik für Dermatologie, Venerologie, Allergologie und Phlebologie Johannes Wesling Klinikum Minden Mühlenkreiskliniken Universitätsklinikum der Ruhr-Universität Bochum
Locations (47):
- Germany (22):
  - Katholisches Klinikum Bochum St. Josef-Hospital, Bochum
  - Elbe Kliniken Stade - Buxtehude GmbH, Buxtehude
  - Klinikum Darmstadt GmbH, Darmstadt
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Helios Klinikum, Erfurt
  - Universitaetsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - SRH Wald-Klinikum, Gera
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Hautklinik Kiel, Kiel
  - Klinikum Ludwigshafen gGmbH, Ludwigshafen
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinik Magdeburg, Magdeburg
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum rechts der Isar, München
  - Fachklinik Muenster-Hornheide, Münster
  - Helios St. Elisabeth Klinik, Oberhausen
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Italy (12):
  - I.R.C.C.S Istituto Tumori "Giovanni Paolo II", Bari
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Toscana Centro - Università di Firenze, Florence
  - Ospedale Policlinico San Martino, Genova
  - ASL1 Avezzano-Sulmona-L'Aquila, L’Aquila
  - Ist. Scien. Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola
  - Forndazione I.R.C.C.S. Istituto nazionale dei tumori, Milan
  - Istituto Tumori Napoli Fondazione G. Pascale, Napoli
  - Università Degli Studi di Napoli Federico II, Napoli
  - AOU Maggiore della Carità - Università del Piemonte Orientale, Novara
  - IDI, Roma
  - Università Cattolica del Sacro Cuore, Roma
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital General Universitari València, Valencia
  - Hospital Universitario La Fe, Valencia
- Switzerland (2):
  - Inselspital, Bern
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Derived] Gutzmer R, Leiter U, Mohr P, Kahler KC, Ascierto PA, Scalvenzi M, Peris K, Perez-Pastor GM, Fernandez-de-Misa R, Botella-Estrada R, Hunger RE, Martelli S, Guneli N, Arntz R, Hauschild A. Interim analysis of the multinational, post-authorization safety study (NISSO) to assess the long-term safety of sonidegib in patients with locally advanced basal cell carcinoma. BMC Cancer. 2024 Nov 14;24(1):1401. doi: 10.1186/s12885-024-13101-z. PMID 39538176